CLINICAL TRIAL: NCT03813030
Title: An Exploratory Study in Healthy Volunteers to Investigate the Cross-talk Between Local Drug Concentrations in the Skin and Systemic Concentrations During Topical Bioequivalence Studies Using Dermal Sampling Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joanneum Research Forschungsgesellschaft mbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: FDA02_AIM4; 2018-002507-33 (EudraCT Number)
Record Dates: First submitted 2019-01-17; First posted 2019-01-23 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2020-07

CONDITIONS: Healthy; Dermal Pharmacokinetic Measurement
Keywords: Dermal open flow microperfusion; Dermal microdialysis
MeSH Terms: interventions — Lidocaine; Prilocaine; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Pilot Study with 6 participants and pivotal study with 20 participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pilot Study (Experimental): Dermal-sampling visit: Measurement of dermal pharmacokinetic (PK) parameter (AUC, Cmax) of lidocaine/ prilocaine using dermal open flow microperfusion (dOFM) and dermal microdialysis (dMD) after topical application of Lidocaine 2.5% and Prilocaine 2.5% cream in 6 participants. Additionally systemic appearance of lidocaine/prilocaine is measured by blood sampling.
  Interventions: Drug: Lidocaine 2.5% and Prilocaine 2.5% cream", USP (2.5% lidocaine, 2.5% prilocaine, Actavis Pharma incorporated, USA); Device: Dermal open flow microperfusion; Device: Dermal Microdialysis; Procedure: Blood sampling in dermal sampling visit
- Pivotal Study (Experimental): Dermal-sampling visit: Measurement of dermal pharmacokinetic (PK) parameter (AUC, Cmax) of lidocaine/ prilocaine using dermal open flow microperfusion (dOFM) and dermal microdialysis (dMD) after topical application of Lidocaine 2.5% and Prilocaine 2.5% cream in 20 participants. Additionally systemic appearance of lidocaine/prilocaine is measured by blood sampling.
  Clearance Visit: Clearance of lidocaine will be evaluated after intravenous infusion of lidocaine.
  Interventions: Procedure: Intravenous infusion of lidocaine; Drug: Lidocaine 2.5% and Prilocaine 2.5% cream", USP (2.5% lidocaine, 2.5% prilocaine, Actavis Pharma incorporated, USA); Drug: Lidocorit 2%-Ampullen" (Gebro Pharma Gesellschaft mit beschränkter Haftung, Austria); Device: Dermal open flow microperfusion; Device: Dermal Microdialysis; Procedure: Blood sampling in dermal sampling visit; Procedure: Blood sampling in clearance visit

INTERVENTIONS:
Procedure: Intravenous infusion of lidocaine — Lidocaine is intravenously administered in clearance visit and blood samples are taken to calculate individual clearance of each participant.
  Arms: Pivotal Study
Drug: Lidocaine 2.5% and Prilocaine 2.5% cream", USP (2.5% lidocaine, 2.5% prilocaine, Actavis Pharma incorporated, USA) — Topical application in dermal-sampling visit
Drug: Lidocorit 2%-Ampullen" (Gebro Pharma Gesellschaft mit beschränkter Haftung, Austria) — Intravenous infusion in clearance visit
  Arms: Pivotal Study
Device: Dermal open flow microperfusion — Dermal open flow microperfusion will be used to collect interstitial fluid in order to assess lidocaine/prilocaine concentration in the dermis.
  Interstitial fluid (ISF) sampling: 1 hour pre-dose and 12 hours post-dose
Device: Dermal Microdialysis — Dermal microdialysis will be used to collect interstitial fluid in order to assess lidocaine/prilocaine concentrations in the dermis.
  Interstitial fluid (ISF) sampling: 1 hour pre-dose and 12 hours post-dose
Procedure: Blood sampling in dermal sampling visit — 1 sample is taken pre-dose and 12 samples are taken post-dose.
Procedure: Blood sampling in clearance visit — 1 sample is taken pre-dose, 3 samples during intravenous infusion and 13 samples post-dose.
  Arms: Pivotal Study

SUMMARY:
This will be a single center, open label, exploratory research study to assess the dermal and systemic PK of marketed products of lidocaine/prilocaine in 26 healthy participants using dermal open flow microperfusion (dOFM) and microdialysis (MD) for dermal sampling.

The clinical study aims to identify potential cross-talk between the extracellular compartments of viable skin and blood circulation during (bioequivalence) BE assessments.

DETAILED DESCRIPTION:
The clinical study is divided into a pilot and a pivotal study.

The pilot study will involve 6 healthy adult participants and in each participant the concentration of lidocaine/prilocaine will be assessed in the dermis and in the systemic circulation after topical application of lidocaine/prilocaine (dermal sampling visit). The pilot study aims to develop the optimal study design for the pivotal study. Thereby the effect of and removal of the topical dose will be tested as well as if this topical dose establishes well quantifiable systemic drug levels that allow an investigation of the cross-talk between skin and systemic circulation within the pivotal study. Further the feasibility of dermal microdialysis (dMD) will be tested and compared with dOFM.

The pivotal study will involve 20 healthy adult participants. It aims to investigate a potential cross-talk between skin and systemic circulation by comparing dermal lidocaine/prilocaine concentrations (assessed with dOFM and MD) and blood lidocaine/prilocaine concentrations in a dermal sampling visit. Furthermore, the systemic clearance of lidocaine will be investigated in each of the 20 participants in a separate clearance visit after intravenous infusion of lidocaine.

In the dermal sampling visits dOFM and microdialysis probes will be inserted into the dermis to monitor the dermal drug concentration up to 12 h post-dose in topically treated as well as untreated skin sites. Blood samples will be drawn to assess the systemic drug levels. All samples will be assayed for lidocaine and prilocaine concentrations. The blood samples in the clearance visit will be assayed for lidocaine only.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult volunteers of age 18 to 65 years (both inclusive).
2. Males or non-pregnant, non-breast feeding females using adequate contraceptive methods or abstinence.
3. Able to read, understand and sign the written informed consent form.
4. Willing to follow the protocol requirements and comply with protocol restrictions.

Exclusion Criteria:

1. Social Habits

   1. Smoker who is not willing to restrain from smoking during the in-house visits.
   2. History of drug and/or alcohol abuse within one year of start of study as judged by the investigator.
2. Medications

   1. Current treatment with systemically effective corticosteroids, monoamine oxidase (MAO) inhibitors, systemic non-selective beta-blockers, warfarin or anticholinergic drugs, or use of any medications referred in the prescription information of the products.
   2. Hormonal contraceptive or hormone replacement therapy, routine vitamins or other prescribed medication are allowed if dose is stable.
3. Diseases

   1. Congenital or idiopathic methemoglobinemia.
   2. History of deep vein thrombosis (DVT)/pulmonary emboly (PE)
   3. Inherited blood disorders (such as factor V Leiden) who are prone to hypercoagulable state
   4. Glucose-6-phosphate dehydrogenase deficiencies
   5. Presence of any acute or chronic diseases or malignancies unless deemed not clinically significant by the investigator.
4. Any reason, which in the opinion of the investigator, would prevent the subject from safely participating in the study.
5. Any abnormalities found at physical examination or vital signs, unless deemed not clinically significant by the investigator.
6. Clinically significant abnormal laboratory evaluation results, as deemed by the investigator.
7. Clinically significant abnormal 12-lead ECG at screening, as deemed by the investigator.
8. Positive results to the test for hepatitis B antigen or hepatitis C antibodies.
9. Positive HIV test.
10. Positive alcohol breath test.
11. Blood donation within 30 days or significant loss of blood or plasma (more than 550 ml) within 90 days prior to screening.
12. Subject who have received an investigational drug within 30 days prior to the initial dose of study medication.
13. Known or suspected allergy/hypersensitivity to lidocaine or prilocaine, known history of sensitivity to local anesthetics of the amide type or to any other component of the product, other related products, or any inactive ingredients.
14. Tattoos or broken and/or damaged skin at the application areas.
15. Active skin diseases like psoriasis or atopic dermatitis, as judged by the investigator.
16. Scarring at the anterior part of the thighs.
17. Subjects prone to keloid or hypertrophic scar formation or any known wound healing disorder.
18. Recent and/or recurrent history of autonomic dysfunction (e.g., recurrent episodes of fainting, palpitations, etc.), as judged by the investigator.
19. Not willing to avoid excessive sun exposure, steam baths, sauna, swimming and other strenuous activities for 14 days after Visit 2 to ensure good tissue regeneration.
20. Not willing to refrain from shaving the planned application sites or using skin care products on the planned application sites for at least 5 days prior to start of Visit 2.
21. Pronounced hairiness on the planned application sites that may negatively affect BE testing.
22. Known allergy/hypersensitivity to any of the materials/supplies used during the study.
23. Presence of needle phobia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Area under the dermal concentration versus time curve for lidocaine (pilot study: 6 participants, pivotal study: 20 participants) | 13 hours
  Dermal concentrations (ng/mL) of lidocaine will be measured to calculate the area under the dermal concentration versus time curve AUC (ng*h/mL).
Area under the dermal concentration time curve for prilocaine (pilot study: 6 participants, pivotal study: 20 participants) | 13 hours
  Dermal concentrations (ng/mL) of prilocaine will be measured to calculate the dermal area under the dermal concentration versus time curve AUC (ng*h/mL).
Maximal dermal concentration of lidocaine (pilot study: 6 participants, pivotal study: 20 participants) | 13 hours
  Dermal concentrations (ng/mL) of lidocaine will be measured to calculate the maximal dermal concentration (ng/mL).
Maximal dermal concentration of prilocaine (pilot study: 6 participants, pivotal study: 20 participants) | 13 hours
  Dermal concentrations (ng/mL) of prilocaine will be measured to calculate the maximal dermal concentration (ng/mL).
Blood lidocaine concentrations versus time curve (pilot study: 6 participants, pivotal study: 20 participants) | 13 hours
  Lidocaine concentrations (ng/mL) in the blood will be measured to obtain the concentration-time curves in the blood.
Blood prilocaine concentrations versus time curve (pilot study: 6 participants, pivotal study: 20 participants) | 13 hours
  Prilocaine concentrations (ng/mL) in the blood will be measured to obtain the concentration-time curves in the blood.

SECONDARY OUTCOMES:
Lidocaine clearance (Pivotal study) - 20 participants | 6 hours post dosing
  Blood concentration (ng/mL) of lidocaine will be measured to obtain the concentration-time curves and to calculated the individual lidocaine clearance (L/min).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pieber, Prof., Principal Investigator — Medical University of Graz
Locations (1):
- Clinical Research Center, Medical University Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bodenlenz M, Tiffner KI, Raml R, Augustin T, Dragatin C, Birngruber T, Schimek D, Schwagerle G, Pieber TR, Raney SG, Kanfer I, Sinner F. Open Flow Microperfusion as a Dermal Pharmacokinetic Approach to Evaluate Topical Bioequivalence. Clin Pharmacokinet. 2017 Jan;56(1):91-98. doi: 10.1007/s40262-016-0442-z. PMID 27539717
- [Background] Bodenlenz M, Dragatin C, Liebenberger L, Tschapeller B, Boulgaropoulos B, Augustin T, Raml R, Gatschelhofer C, Wagner N, Benkali K, Rony F, Pieber T, Sinner F. Kinetics of Clobetasol-17-Propionate in Psoriatic Lesional and Non-Lesional Skin Assessed by Dermal Open Flow Microperfusion with Time and Space Resolution. Pharm Res. 2016 Sep;33(9):2229-38. doi: 10.1007/s11095-016-1960-y. Epub 2016 Jun 6. PMID 27271272
- [Background] Rowland M, Thomson PD, Guichard A, Melmon KL. Disposition kinetics of lidocaine in normal subjects. Ann N Y Acad Sci. 1971 Jul 6;179:383-98. doi: 10.1111/j.1749-6632.1971.tb46915.x. No abstract available. PMID 5285383
- [Background] Benfeldt E, Hansen SH, Volund A, Menne T, Shah VP. Bioequivalence of topical formulations in humans: evaluation by dermal microdialysis sampling and the dermatopharmacokinetic method. J Invest Dermatol. 2007 Jan;127(1):170-8. doi: 10.1038/sj.jid.5700495. Epub 2006 Jul 27. PMID 16874309
- [Background] Estebe JP. Intravenous lidocaine. Best Pract Res Clin Anaesthesiol. 2017 Dec;31(4):513-521. doi: 10.1016/j.bpa.2017.05.005. Epub 2017 May 30. PMID 29739540